CLINICAL TRIAL: NCT01651663
Title: Double-blind, Randomized, Placebo-controlled Clinical Study Investigating Efficacy and Safety of Arbidol (Umifenovir) in Treatment and Prophylaxis of Influenza and Common Cold.
Brief Title: A Study of Arbidol (Umifenovir) for Treatment and Prophylaxis of Influenza and Common Cold
Acronym: ARBITR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmstandard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARB-M1/P01-11
Record Dates: First submitted 2012-07-02; First posted 2012-07-27 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — umifenovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arbidol (Umifenovir) (Experimental)
  Interventions: Drug: Arbidol (Umifenovir)
- placebo (Placebo Comparator)
  Interventions: Other: placebo
- Arbidol (Umifenovir) prophylaxis (Experimental)
  Interventions: Drug: Arbidol (Umifenovir)
- placebo prophylaxis (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Arbidol (Umifenovir) — Arbidol (Umifenovir)/Placebo will be administered at a dosage of 800 mg/day (2 capsules q.i.d.) for 5 days.
  Arms: Arbidol (Umifenovir)
Other: placebo — Arbidol (Umifenovir)/Placebo will be administered at a dosage of 800 mg/day (2 capsules q.i.d.) for 5 days.
  Arms: placebo
Drug: Arbidol (Umifenovir) — Medically healthy exposed subjects will be administered Arbidol (Umifenovir)/Placebo at a dosage of 200 mg/day (2 capsules q.d.) for 10 days.
  Arms: Arbidol (Umifenovir) prophylaxis
Other: placebo — Medically healthy exposed subjects will be administered Arbidol (Umifenovir)/Placebo at a dosage of 200 mg/day (2 capsules q.d.) for 10 days.
  Arms: placebo prophylaxis

SUMMARY:
The purpose of this study is to determine whether Arbidol (Umifenovir) is effective in the treatment and Prophylaxis of Influenza and Common Cold

DETAILED DESCRIPTION:
Influenza virus infections result in major health and economic burdens worldwide. The World Health Organization estimates that the average global burden of interpandemic influenza is approximately 1 billion cases of influenza, from 3 to 5 million cases of severe illness, and from 300 000 to 500 000 deaths annually. Arbidol (Umifenovir) is currently licensed for the treatment and prevention of influenza in Russian Federation. Arbidol (Umifenovir) has a direct antiviral effect. Arbidol (Umifenovir) belongs to fusion inhibitors; it interacts with the virus hemagglutinin and thus prevents fusion of the viral envelope with cell membranes. The aim of the study is to obtain additional data on safety and therapeutic efficacy of investigational product Arbidol (Umifenovir) in patients with a diagnosis of influenza and common cold. Furthermore, study of viral resistance in patients with seasonal influenza infection treated with Arbidol (Umifenovir) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Signed Patient Information and Informed Consent Form.
* Male and female patients from 18 to 65 years.
* Out-patients with uncomplicated* form of common cold or influenza.
* Illness duration no more than 36 hours.
* At least one episode of body temperature 38°C or higher during the past 36 hours.
* Presence of at least one of the following symptoms: Headache, fatigue/malaise, pain/aches in muscles, fever/chills.
* Patient's ability to adequately cooperate.

Exclusion Criteria:

* A history of allergic reactions to the investigational drug Arbidol (Umifenovir) or hypersensitivity to the drug.
* Illness duration over 36 hours.
* Any complications of influenza/common cold or signs of severe or progressive disease* at the moment of selection for participation in the study.
* A history of influenza vaccination carried out in the last 12 months.
* Evidence of severe hematological, immunological, pulmonary, urogenital, gastrointestinal, hepatic, renal, endocrine, metabolic, psychiatric, dermatovenereological diseases, collagenoses, nutritional disorders, which are known from patient's history, physical examination or laboratory tests, that may limit the patient from participating in the study or which may affect the results of the study.
* Participation in other clinical studies in the past 4 months.
* Common cold or other infection during last 4 weeks before enrollment.
* Administration of Arbidol (Umifenovir) during last 4 weeks before the onset of disease.
* Administration of immunomodulators, interferon inducers, homeopathic, hormonal, antiviral and antibacterial drugs during last 4 weeks before the selection for participation in the study.
* Alcohol or substance abuse.
* Hospitalization at the moment of selection for participation in the study.
* Pregnant or lactating women.
* Any other associated disease or condition which, in the opinion of the investigator, might restrict or impede the patient's participation in the study or affect the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Duration of clinical illness among patients with common cold and influenza treated with Arbidol vs placebo. | Baseline up to 20 days
Time to alleviation of influenza and common cold clinical symptoms | Baseline up to 20 days
Number of Adverse Events that are probably or definitely related to Arbidol | Baseline up to 20 days

SECONDARY OUTCOMES:
Number of clinical complications associated with influenza and common cold among treatment group vs placebo | Baseline up to 20 days
The time to no detectable influenza virus by culture for the throat and nose swabs, assessed by PCR | Day 3, Day 4, Day 5, Day 6, Day 7, Day 8
Occurrence of influenza and common cold among participants in prophylaxis group diagnosed by physician according to history and physical examination and laboratory tests if was necessary | Baseline up to 20 days
Frequency of emergence of antiviral resistance | Baseline up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Kiselev, Dr.Biol.Sci., Principal Investigator — Research Instituete of Influenza
Locations (2):
- Russia (2):
  - Research Institute of Influenza, Saint Petersburg
  - Saratov